CLINICAL TRIAL: NCT04033068
Title: Observer Blinded, Randomized Trial to Evaluate Safety and Immunogenicity of a Novel Vaccine Formulation MV-ZIKA-RSP
Brief Title: Safety and Immunogenicity of a Novel Vaccine Formulation MV-ZIKA-RSP (V187-001)
Acronym: MV-ZIKA-RSP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V187-001; 2019-000840-93 (EudraCT Number); MV-ZIKA-RSP (Other: Themisbio)
Record Dates: First submitted 2019-07-08; First posted 2019-07-25 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: Zika Virus Infection
Keywords: Zika virus; mosquito-borne pathogen; Zika fever
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Two MV-ZIKA-RSP vaccinations (high dose) (Experimental): 14 Participants will receive MV-ZIKA-RSP 1 x10E5/dose on day 0 and day 28
  Interventions: Biological: Two MV-ZIKA-RSP vaccinations (high dose)
- Two MV-ZIKA-RSP vaccination (low dose) (Experimental): 14 Participants will receive MV-ZIKA-RSP 2,5 x10E4 /dose on day 0 and day 28
  Interventions: Biological: Two MV-ZIKA-RSP vaccination (low dose)
- One MV-ZIKA-RSP vaccination (high dose) and one placebo (Experimental): 12 Participants will receive MV-ZIKA-RSP 1 x10E5/dose on day 0 and placebo on day 28
  Interventions: Biological: One MV-ZIKA-RSP vaccination (high dose) and one placebo
- Two placebo injection (Placebo Comparator): 8 Participants will receive placebo on day 0 and placebo on day 28
  Interventions: Other: Two placebo injection

INTERVENTIONS:
Biological: Two MV-ZIKA-RSP vaccinations (high dose) — In this arm of the study, 14 participants will receive:
  1. V1= day 0; dose vaccination with MV-ZIKA-RSP (high dose).
  2. V2= day 28; dose vaccination with MV-ZIKA-RSP (high dose).
  Description:
  Visit 1: Participants will receive their first vaccination with MV-ZIKA-RSP (high dose) Visit 2: Participants will receive their second vaccination with MV-ZIKA-RSP (high dose)
  Arms: Two MV-ZIKA-RSP vaccinations (high dose)
Biological: Two MV-ZIKA-RSP vaccination (low dose) — In this arm of the study, 14 participants will receive:
  1. V1= day 0; dose vaccination with MV-ZIKA-RSP (low dose).
  2. V2= day 28; dose vaccination with MV-ZIKA-RSP (low dose).
  Description:
  Visit 1: Participants will receive their first vaccination with MV-ZIKA-RSP (low dose) Visit 2: Participants will receive their second vaccination with MV-ZIKA-RSP (low dose)
  Arms: Two MV-ZIKA-RSP vaccination (low dose)
Biological: One MV-ZIKA-RSP vaccination (high dose) and one placebo — In this arm of the study, 12 participants will receive:
  1. V1= day 0; dose vaccination with MV-ZIKA-RSP (high dose).
  2. V2= day 28; treatment with placebo
  Description:
  Visit 1: Participants will receive their first vaccination with MV-ZIKA-RSP (high dose) Visit 2: Participants will receive their second treatment with placebo
  Arms: One MV-ZIKA-RSP vaccination (high dose) and one placebo
Other: Two placebo injection — In this arm of the study, 8 participants will receive:
  1. V1= day 0; placebo treatment
  2. V2= day 28; placebo treatment
  Description:
  Visit 1: Participants will receive their first treatment with placebo Visit 2: Participants will receive their second treatment with placebo
  Other Names: Placebo arm
  Arms: Two placebo injection

SUMMARY:
This study is designed to investigate, at first, safety and tolerability of a novel liquid vaccine formulation named MV-ZIKA-RSP, in healthy adults aged 18 to 55 years

DETAILED DESCRIPTION:
This is an observer-blinded, block-randomized, dose-finding, phase I trial, comparing different dose levels of MV-ZIKA-RSP to evaluate the safety, tolerability, and immunogenicity, of this novel ZIKA-RSP vaccine. Placebo (physiological saline solution) will be applied to blind the different treatment schedules.

After the screening procedures, 48 healthy male and female volunteers aged 18-55 years will be randomly assigned to one of four treatment groups (A, B, C or D). Participants will be assessed for immunogenicity on days 0, 28 and 56 (treatment period), as confirmed by the presence of functional anti-zika-rsp antibodies determined by (PRNT50) and by ELISA, at the same time safety will be also assessed. After the treatment period, participants will be called by phone (day 182) for evaluation of safety follow-up.

The investigator and site personnel assessing AEs, all participants, as well as one of the sponsor's representatives involved in the monitoring and conduct of the study will be blinded to which vaccine was administered. Only the unblinded monitor, site personnel performing randomization, preparation and administration of IMP will be unblinded.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any trial-related activities
2. Healthy men or women aged 18 to 55 years on the day of consenting
3. Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the investigator and to comply with the requirements of the entire study
4. All female participants must have a negative urine pregnancy serum pregnancy test at screening
5. Willingness not to become pregnant or to father a child during the entire study period by practising reliable methods of contraception as specified in protocol section 8.11.4
6. Availability during the duration of the trial
7. Normal findings in medical history and physical examination or the investigator considers all abnormalities to be clinically irrelevant
8. Normal laboratory values or the investigator considers all abnormalities to be clinically irrelevant (unless otherwise specified in exclusion criteria)

Exclusion Criteria:

1. Participation in another clinical study (including exposure to an investigational medicinal product or device) within one month before the screening visit or planned concurrent participation in another clinical study before completion of the treatment period (day 56)
2. History of immunodeficiency, known human immunodeficiency virus (HIV) infection or current hepatitis B/C infection
3. Strong anamnestic evidence for or confirmed the history of or current infection with Zika- or Dengue-virus
4. History of drug addiction including alcohol dependence within the last 2 years
5. Inability or unwillingness to avoid intake of more than around 20g alcohol per day during 48 hours after each vaccination (equals roughly 0.5 L beer or 0.25 L of wine)
6. Vaccination within 4 weeks prior to first vaccination or planning to receive any non-study vaccine until the end of the treatment period (day 56)
7. Prior receipt of any Zika or Chikungunya vaccine
8. History of moderate or severe arthritis or arthralgia within the past 3 months prior to Screening Visit
9. Recent infection within 1 week prior to Screening Visit (possibility of deferral)
10. Blood donations including plasma donations, 90 days prior to Screening Visit and anticipated blood, plasma, tissue, sperm or organ donation, throughout the study until the end of the treatment period (day 56)
11. Clinically relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, inflammatory, autoimmune or neurological diseases or clinically relevant abnormal laboratory values, that in the opinion of the investigator may interfere with the aim of the study
12. History of neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) within the past 5 years or a history of any haematological malignancy
13. Behavioural, cognitive, or psychiatric condition that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
14. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the vaccine
15. History of anaphylaxis to drugs or other allergic reactions, which the investigator considers compromising the safety of the volunteer
16. Abnormal laboratory values which, at the discretion of the investigator should lead to the exclusion of the subject
17. Use of medication during 2 weeks before the first vaccination and throughout the study, which the investigator considers affecting the validity of the study, except hormonal contraception or hormonal replacement therapy in female participants. (Prior to taking any medication within 72 h before study vaccination, the subject should consult the investigator)
18. Use of immunosuppressive drugs like corticosteroids (excluding topical preparations) within 30 days prior to first IMP administration, or anticipated use until completion of the end of treatment visit Receipt of blood products or immunoglobulins within 120 days prior to the Screening Visit or anticipated receipt of any blood product or immunoglobulin before completion of the treatment period (day 56)
19. Pregnancy (positive pregnancy test at screening or during the treatment period) or lactation at screening, or planning to become pregnant during the treatment period
20. Unreliable contraception methods (for details please refer to protocol section 8.11.4)
21. Persons in a direct relationship with the sponsor, an investigator or other study team members. Direct dependent relationships include close relatives (i.e. children, parents, partner/spouse, siblings) as well as employees of the study site or the sponsor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Institute of Specific Prophylaxis and Tropical Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rossi SL, Comer JE, Wang E, Azar SR, Lawrence WS, Plante JA, Ramsauer K, Schrauf S, Weaver SC. Immunogenicity and Efficacy of a Measles Virus-Vectored Chikungunya Vaccine in Nonhuman Primates. J Infect Dis. 2019 Jul 31;220(5):735-742. doi: 10.1093/infdis/jiz202. PMID 31053842
- See also: Sponsor Web Page — http://www.themis.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened within two weeks prior to randomization.
Groups:
- Group A: V187 (High Dose) - V187 (High Dose): Participants receive V187 at a high dose of 1x10^5 Tissue Culture Infective Dose 50% (TCID50) on Day 0 (first dose) and Day 28 (second dose) via intramuscular (IM) injection.
- Group B: V187 (Low Dose) - V187 (Low Dose): Participants receive V187 at a low dose of 2.5x10^4 TCID50 on Day 0 (first dose) and Day 28 (second dose) via IM injection.
- Group C: V187 (High Dose) - Placebo: Participants receive V187 at a high dose of 1x10^5 TCID50 on Day 0 (first dose) and V187-matching placebo on Day 28 (second dose) via IM injection.
- Group D: Placebo - Placebo: Participants receive V187-matching placebo on Day 0 (first dose) and Day 28 (second dose) via IM injection.
Period: Overall Study
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Started | 14 | 14 | 12 | 8
First Dose | 14 | 14 | 12 | 8
Second Dose | 14 | 14 | 11 | 7
Completed | 14 | 13 | 11 | 7
Not Completed | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Inclusion / exclusion criteria not fulfilled | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo | Total
Number analyzed (Participants) | 14 | 14 | 12 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (9.15) | 35.5 (10.09) | 33.4 (10.74) | 39.3 (12.41) | 36.5 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 9 | 3 | 31
  Male | 4 | 5 | 3 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 14 | 14 | 12 | 7 | 47
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE) up to Day 56
Description: An AE is any untoward medical occurrence in a participant to whom an investigational medicinal product has been administered, not necessarily caused by or related to that product. As specified by the protocol, the percentage of participants who experience an AE up to study Day 56 was presented.
Time Frame: Up to Day 56
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Percentage of Participants | 92.9 | 92.9 | 91.7 | 62.5
Statistical Analysis 1: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Test type: Superiority; p = 0.2003, Fisher-Freeman-Halton Test

2. Secondary Outcome: Percentage of Participants Who Experienced a Solicited AE up to Day 182
Description: An AE is any untoward medical occurrence in a participant to whom an investigational medicinal product has been administered, not necessarily caused by or related to that product. Solicited AEs include local solicited AEs (e.g. injection site pain, tenderness, erythema/redness, swelling, itching and induration) and systemic solicited AEs (e.g. nausea, vomiting, arthralgia, headache, fatigue, myalgia, fever, pain in limb, rash and flu-like symptoms). Solicited AEs were recorded in a diary by the participant and verified by the investigator. As specified by the protocol, the percentage of participants who experience a solicited AE up to study Day 182 was presented.
Time Frame: Up to Day 182
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Percentage of Participants | 92.9 | 78.6 | 83.3 | 50.0
Statistical Analysis 1: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Test type: Superiority; p = 0.1448, Fisher-Freeman-Halton Test

3. Secondary Outcome: Percentage of Participants Who Experienced an Unsolicited AE up to Day 182
Description: An AE is any untoward medical occurrence in a participant to whom an investigational medicinal product has been administered, not necessarily caused by or related to that product. Unsolicited or spontaneous AEs were recorded in a diary by the participant and verified by the investigator. As specified by the protocol, the percentage of participants who experienced an unsolicited AE up to study Day 182 was presented.
Time Frame: Up to Day 182
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Percentage of Participants | 57.1 | 71.4 | 58.3 | 62.5
Statistical Analysis 1: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Test type: Superiority; p = 0.9111, Fisher-Freeman-Halton Test

4. Secondary Outcome: Percentage of Participants Who Experienced a Serious Adverse Event (SAE) up to Day 182
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect or is another important medical event deemed as much by medical or scientific judgement. As specified by the protocol, the percentage of participants who experience an SAE up to study Day 182 was presented.
Time Frame: Up to Day 182
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Percentage of Participants | 0.0 | 7.1 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Test type: Superiority; p = 1.0000, Fisher-Freeman-Halton Test

5. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-ZIKA-RSP (Zikavirus Recombinant Subviral Particle) Antibodies by Virus Neutralization Test (VNT) on Days 0, 28 and 56
Description: The induction of functional anti-ZIKA-RSP antibodies by V187 was investigated in sera from participants by means of a VNT, an immunoassay that detects and quantifies antibodies in serum samples that can neutralize infectious Zika virions. As specified by the protocol, the GMT of anti-ZIKA-RSP antibodies by the VNT on Day 0 (first dose), Day 28 (second dose) and Day 56 (follow-up assessment) was presented. Values below the lower limit of quantification (LLOQ) were set to the half of the true LLOQ value and values above the upper limit of quantification (ULOQ) were set to the true ULOQ value for calculations.
Time Frame: Day 0, Day 28 and Day 56
Population: All randomized participants without protocol deviations that could impact immune response, who had anti-ZIKA-RSP antibody VNT data available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 12 | 13 | 10 | 7
Titers
  Day 0 | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0]
  Day 28 | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0]
  Day 56 | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0] | 10.0 (10.0) [10.0 to 10.0]

6. Secondary Outcome: GMT of Anti-ZIKA-RSP Antibodies by Enzyme Linked Immunosorbent Assay (ELISA) on Days 0, 28 and 56
Description: The induction of functional anti-ZIKA-RSP antibodies by V187 was investigated in sera from participants by means of Immunoglobulin G (IgG) ELISA, an immunoassay that quantifies anti-ZIKA-RSP IgG. As specified by the protocol, the GMT of anti-ZIKA-RSP antibodies by ELISA on Day 0 (first dose), Day 28 (second dose) and Day 56 (follow-up assessment) was presented. Values below the LLOQ were set to the half of the true LLOQ value and values above the ULOQ were set to the true ULOQ value for calculations.
Time Frame: Day 0, Day 28 and Day 56
Population: All randomized participants without protocol deviations that could impact immune response, who had anti-ZIKA-RSP antibody ELISA data available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 12 | 13 | 10 | 7
Titers
  Day 0 | 2107.0 (579.6) [579.6 to 7659.7] | 2310.9 (829.1) [829.1 to 6440.8] | 2780.8 (1269.3) [1269.3 to 6092.5] | 1759.2 (408.9) [408.9 to 7568.2]
  Day 28 | 4084.2 (1348.4) [1348.4 to 12370.5] | 3529.3 (1570.9) [1570.9 to 7929.5] | 4219.7 (2008.3) [2008.3 to 8866.3] | 1821.1 (421.3) [421.3 to 7872.4]
  Day 56 | 5908.4 (2210.4) [2210.4 to 15792.8] | 4600.6 (2386.1) [2386.1 to 8870.4] | 3485.9 (1783.3) [1783.3 to 6813.9] | 2059.0 (435.5) [435.5 to 9734.7]
Statistical Analysis 1: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose); Day 0; Test type: Superiority; p = 0.9990, ANOVA; GMT Ratio = 0.9, 95% CI 2-sided [0.2 to 5.5]
Statistical Analysis 2: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group C: V187 (High Dose) - Placebo; Day 0; Test type: Superiority; p = 0.9798, ANOVA; GMT Ratio = 0.8, 95% CI 2-sided [0.1 to 5.2]
Statistical Analysis 3: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group D: Placebo - Placebo; Day 0; Test type: Superiority; p = 0.9958, ANOVA; GMT Ratio = 1.2, 95% CI 2-sided [0.1 to 10.1]
Statistical Analysis 4: Comparison: Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo; Day 0; Test type: Superiority; p = 0.9935, ANOVA; GMT Ratio = 0.8, 95% CI 2-sided [0.1 to 5.5]
Statistical Analysis 5: Comparison: Group B: V187 (Low Dose) - V187 (Low Dose) vs Group D: Placebo - Placebo; Day 0; Test type: Superiority; p = 0.9852, ANOVA; GMT Ratio = 1.3, 95% CI 2-sided [0.2 to 10.7]
Statistical Analysis 6: Comparison: Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Day 0; Test type: Superiority; p = 0.9440, ANOVA; GMT Ratio = 1.6, 95% CI 2-sided [0.2 to 14.4]
Statistical Analysis 7: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose); Day 28; Test type: Superiority; p = 0.9943, ANOVA; GMT Ratio = 1.2, 95% CI 2-sided [0.2 to 5.5]
Statistical Analysis 8: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group C: V187 (High Dose) - Placebo; Day 28; Test type: Superiority; p = 0.9999, ANOVA; GMT Ratio = 1.0, 95% CI 2-sided [0.2 to 5.1]
Statistical Analysis 9: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group D: Placebo - Placebo; Day 28; Test type: Superiority; p = 0.6476, ANOVA; GMT Ratio = 2.2, 95% CI 2-sided [0.4 to 14.3]
Statistical Analysis 10: Comparison: Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo; Day 28; Test type: Superiority; p = 0.9911, ANOVA; GMT Ratio = 0.8, 95% CI 2-sided [0.2 to 4.3]
Statistical Analysis 11: Comparison: Group B: V187 (Low Dose) - V187 (Low Dose) vs Group D: Placebo - Placebo; Day 28; Test type: Superiority; p = 0.7647, ANOVA; GMT Ratio = 1.9, 95% CI 2-sided [0.3 to 12.0]
Statistical Analysis 12: Comparison: Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Day 28; Test type: Superiority; p = 0.6447, ANOVA; GMT Ratio = 2.3, 95% CI 2-sided [0.3 to 15.8]
Statistical Analysis 13: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group B: V187 (Low Dose) - V187 (Low Dose); Day 56; Test type: Superiority; p = 0.9638, ANOVA; GMT Ratio = 1.3, 95% CI 2-sided [0.3 to 5.3]
Statistical Analysis 14: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group C: V187 (High Dose) - Placebo; Day 56; Test type: Superiority; p = 0.7837, ANOVA; GMT Ratio = 1.7, 95% CI 2-sided [0.4 to 7.7]
Statistical Analysis 15: Comparison: Group A: V187 (High Dose) - V187 (High Dose) vs Group D: Placebo - Placebo; Day 56; Test type: Superiority; p = 0.3427, ANOVA; GMT Ratio = 2.9, 95% CI 2-sided [0.5 to 15.3]
Statistical Analysis 16: Comparison: Group B: V187 (Low Dose) - V187 (Low Dose) vs Group C: V187 (High Dose) - Placebo; Day 56; Test type: Superiority; p = 0.9578, ANOVA; GMT Ratio = 1.3, 95% CI 2-sided [0.3 to 5.8]
Statistical Analysis 17: Comparison: Group B: V187 (Low Dose) - V187 (Low Dose) vs Group D: Placebo - Placebo; Day 56; Test type: Superiority; p = 0.5637, ANOVA; GMT Ratio = 2.2, 95% CI 2-sided [0.4 to 11.7]
Statistical Analysis 18: Comparison: Group C: V187 (High Dose) - Placebo vs Group D: Placebo - Placebo; Day 56; Test type: Superiority; p = 0.8471, ANOVA; GMT Ratio = 1.7, 95% CI 2-sided [0.3 to 9.6]

7. Secondary Outcome: T-Cell Immune Response Assessed by Number of Spot Forming Cells (SFC) Per Million Peripheral Blood Mononuclear Cells (PBMCs) Measured by Interferon (IFN)-γ Enzyme-linked Immune Adsorbent Spot (ELISpot) Assay on Day 56
Description: Immune response mediated by functional T-cells was investigated using an IFNγ enzyme-linked immune adsorbent spot (ELISpot) assay. This is an immunoassay that quantifies IFNγ producing cells by assessing the number of SFCs per 10^6 PBMCs stimulated with a peptide pool containing the viral protein prM*; a precipitate forms and appears as spots at the sites of cytokine localization, with each individual spot representing an individual cytokine-secreting cell. As specified by the protocol, median of the number of IFNγ SFCs per 10^6 PBMCs on Day 56 was presented. Values below the LLOQ were set to the half of the true LLOQ value and values above the ULOQ were set to the true ULOQ value for calculations.
Time Frame: Day 56
Population: All randomized participants without protocol deviations that could impact immune response, who had IFNγ SFC data available.
Measure: Median (Inter-Quartile Range); unit: SFC/10^6 PBMC
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 12 | 13 | 10 | 7
SFC/10^6 PBMC | 0.0 (0.0) [0.0 to 9.0] | 0.0 (0.0) [0.0 to 6.0] | 10.0 (3.0) [3.0 to 30.0] | 2.5 (1.0) [1.0 to 10.5]

8. Secondary Outcome: T-Cell Immune Response Assessed by Number of SFC Per Million PBMCs Measured by Interleukin-2 (IL-2) ELISpot Assay on Day 56
Description: Immune response mediated by functional T-cells was investigated using an IL-2 ELISpot assay. This is an immunoassay that quantifies IL-2 producing cells by assessing the number of SFCs per 10^6 PBMCs stimulated with a peptide pool containing the viral protein prM*; a precipitate forms and appears as spots at the sites of cytokine localization, with each individual spot representing an individual cytokine-secreting cell. As specified by the protocol, median of the number of IL-2 SFCs per 10^6 PBMCs on Day 56 was presented. Values below the LLOQ were set to the half of the true LLOQ value and values above the ULOQ were set to the true ULOQ value for calculations.
Time Frame: Day 56
Population: All randomized participants without protocol deviations that could impact immune response, who had IL-2 SFC data available.
Measure: Median (Inter-Quartile Range); unit: SFC/10^6 PBMC
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 12 | 13 | 10 | 7
SFC/10^6 PBMC | 7.5 (0.0) [0.0 to 15.5] | 0.0 (0.0) [0.0 to 18.0] | 0.0 (0.0) [0.0 to 5.0] | 1.0 (0.0) [0.0 to 3.0]

9. Secondary Outcome: Laboratory Parameters (Hematology): Concentration of Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets on Days 28 and 56
Description: Hematological parameters were investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available hematology data.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Giga cells per liter
  Basophils Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Basophils Day 28 | 0.05 (0.05) | 0.06 (0.06) | 0.03 (0.05) | 0.06 (0.05)
  Basophils Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Basophils Day 56 | 0.04 (0.05) | 0.07 (0.06) | 0.02 (0.04) | 0.07 (0.05)
  Eosinophils Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Eosinophils Day 28 | 0.19 (0.12) | 0.17 (0.14) | 0.15 (0.12) | 0.17 (0.14)
  Eosinophils Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Eosinophils Day 56 | 0.20 (0.13) | 0.16 (0.13) | 0.13 (0.13) | 0.16 (0.08)
  Leukocytes Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Leukocytes Day 28 | 7.11 (1.30) | 7.47 (3.82) | 5.51 (1.58) | 7.49 (2.96)
  Leukocytes Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Leukocytes Day 56 | 6.81 (1.56) | 7.21 (2.58) | 5.55 (1.48) | 7.83 (3.53)
  Lymphocytes Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Lymphocytes Day 28 | 2.01 (0.57) | 1.99 (0.77) | 1.74 (0.43) | 2.03 (0.93)
  Lymphocytes Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Lymphocytes Day 56 | 1.94 (0.39) | 1.96 (0.83) | 1.76 (0.44) | 1.85 (1.02)
  Monocytes Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Monocytes Day 28 | 0.54 (0.10) | 0.52 (0.13) | 0.45 (0.10) | 0.49 (0.22)
  Monocytes Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Monocytes Day 56 | 0.51 (0.09) | 0.51 (0.11) | 0.43 (0.12) | 0.52 (0.17)
  Neutrophils Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Neutrophils Day 28 | 4.29 (1.02) | 4.74 (3.09) | 3.15 (1.21) | 4.73 (2.22)
  Neutrophils Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Neutrophils Day 56 | 4.11 (1.39) | 4.49 (1.72) | 3.20 (1.12) | 5.28 (2.68)
  Platelets Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Platelets Day 28 | 275.0 (82.43) | 290.93 (74.22) | 236.45 (45.65) | 274.86 (60.78)
  Platelets Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Platelets Day 56 | 273.21 (73.62) | 286.93 (75.68) | 229.55 (47.98) | 281.17 (60.50)

10. Secondary Outcome: Laboratory Parameter (Hematology): Concentration of Erythrocytes on Days 28 and 56
Description: Hematological parameters were investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of erythrocytes on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available hematology data.
Measure: Mean (Standard Deviation); unit: Trillions of cells per liter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Trillions of cells per liter
  Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 28 | 4.73 (0.44) | 4.49 (0.49) | 4.59 (0.19) | 4.80 (0.42)
  Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Day 56 | 4.67 (0.40) | 4.56 (0.44) | 4.63 (0.23) | 4.83 (0.62)

11. Secondary Outcome: Laboratory Parameter (Hematology): Concentration of Hematocrit on Days 28 and 56
Description: Hematological parameters were investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of hematocrit on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available hematology data.
Measure: Mean (Standard Deviation); unit: Liter of cells per liter of blood
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Liter of cells per liter of blood
  Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 28 | 0.41 (0.03) | 0.39 (0.05) | 0.40 (0.02) | 0.43 (0.03)
  Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Day 56 | 0.41 (0.03) | 0.40 (0.05) | 0.41 (0.02) | 0.43 (0.05)

12. Secondary Outcome: Laboratory Parameter (Hematology): Concentration of Hemoglobin on Days 28 and 56
Description: Hematological parameters were investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of hemoglobin on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available hematology data.
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Grams per deciliter
  Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 28 | 14.06 (1.09) | 13.57 (2.11) | 13.82 (0.70) | 14.63 (1.19)
  Day 56: number analyzed (Participants) | 14 | 14 | 11 | 6
  Day 56 | 13.89 (1.02) | 13.64 (2.00) | 13.79 (0.74) | 14.63 (1.60)

13. Secondary Outcome: Laboratory Parameters (Clinical Chemistry): Concentration of Alanine Aminotransferase, Alkaline Phosphatase and Aspartate Aminotransferase on Days 28 and 56
Description: Clinical chemistry parameters were investigated in sera from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of alanine aminotransferase, alkaline phosphatase and aspartate aminotransferase on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available clinical chemistry data.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Units per liter
  Alanine Aminotransferase Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Alanine Aminotransferase Day 28 | 35.00 (21.91) | 20.14 (8.79) | 21.09 (7.38) | 26.00 (13.66)
  Alanine Aminotransferase Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Alanine Aminotransferase Day 56 | 35.21 (19.86) | 22.29 (13.75) | 22.18 (8.32) | 22.14 (8.36)
  Alkaline Phosphatase Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Alkaline Phosphatase Day 28 | 65.29 (14.62) | 63.43 (20.63) | 63.18 (16.14) | 79.86 (23.36)
  Alkaline Phosphatase Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Alkaline Phosphatase Day 56 | 65.50 (15.81) | 65.14 (20.72) | 59.73 (16.63) | 77.43 (23.78)
  Aspartate Aminotransferase Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Aspartate Aminotransferase Day 28 | 29.21 (19.26) | 21.64 (6.45) | 22.36 (3.29) | 24.57 (8.04)
  Aspartate Aminotransferase Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Aspartate Aminotransferase Day 56 | 29.43 (12.02) | 19.36 (5.47) | 22.55 (4.32) | 23.71 (6.26)

14. Secondary Outcome: Laboratory Parameters (Clinical Chemistry): Concentration of Sodium, Calcium and Potassium on Days 28 and 56
Description: Clinical chemistry parameters were investigated in sera from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of sodium, calcium and potassium on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available clinical chemistry data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Millimoles per liter
  Sodium Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Sodium Day 28 | 139.57 (1.65) | 139.5 (1.95) | 139.82 (1.78) | 141.43 (1.62)
  Sodium Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Sodium Day 56 | 139.64 (1.95) | 139.86 (2.07) | 139.45 (2.02) | 140.29 (1.80)
  Calcium Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Calcium Day 28 | 2.39 (0.08) | 2.37 (0.08) | 2.36 (0.09) | 2.40 (0.08)
  Calcium Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Calcium Day 56 | 2.38 (0.09) | 2.36 (0.09) | 2.36 (0.08) | 2.34 (0.08)
  Potassium Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Potassium Day 28 | 4.72 (0.44) | 4.63 (0.34) | 4.35 (0.29) | 4.53 (0.26)
  Potassium Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Potassium Day 56 | 4.61 (0.47) | 4.58 (0.42) | 4.67 (0.54) | 4.70 (0.30)

15. Secondary Outcome: Laboratory Parameters (Clinical Chemistry): Concentration of Bilirubin and Creatinine on Days 28 and 56
Description: Clinical chemistry parameters were investigated in sera from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the concentration of bilirubin and creatinine on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available clinical chemistry data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
milligrams per deciliter
  Bilirubin Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Bilirubin Day 28 | 0.40 (0.22) | 0.39 (0.27) | 0.44 (0.16) | 0.50 (0.35)
  Bilirubin Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Bilirubin Day 56 | 0.42 (0.13) | 0.41 (0.24) | 0.42 (0.13) | 0.46 (0.19)
  Creatinine Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Creatinine Day 28 | 0.83 (0.18) | 0.71 (0.15) | 0.77 (0.13) | 0.84 (0.13)
  Creatinine Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Creatinine Day 56 | 0.82 (0.13) | 0.76 (0.13) | 0.79 (0.12) | 0.81 (0.17)

16. Secondary Outcome: Laboratory Parameter (Urinalysis): pH on Days 28 and 56
Description: Urinalysis parameters were investigated in urine samples from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the pH on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available urinalysis data.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
pH
  Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 28 | 5.79 (1.05) | 5.43 (0.65) | 5.82 (0.60) | 5.57 (0.79)
  Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 56 | 5.71 (1.07) | 5.79 (0.89) | 5.82 (0.87) | 5.14 (0.38)

17. Secondary Outcome: Laboratory Parameter (Urinalysis): Specific Gravity on Days 28 and 56
Description: Urinalysis parameters were investigated in urine samples from participants by means of clinical laboratory assays and evaluated by the investigator. As specified by the protocol, the specific gravity on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available urinalysis data.
Measure: Mean (Standard Deviation); unit: grams per milliliter
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
grams per milliliter
  Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 28 | 1.014 (0.005) | 1.011 (0.007) | 1.010 (0.008) | 1.011 (0.009)
  Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Day 56 | 1.013 (0.009) | 1.012 (0.007) | 1.013 (0.004) | 1.009 (0.005)

18. Secondary Outcome: Laboratory Parameters (Urinalysis): Percentage of Participants Negative for Bilirubin, Erythrocytes, Ketones, Leukocytes, Nitrite and Protein on Days 28 and 56
Description: Urinalysis parameters were investigated in urine samples from participants by means of clinical laboratory assays and evaluated by the investigator. Bilirubin, erythrocytes, ketones, leukocytes, nitrite and protein levels were defined as negative by the local laboratory and reported at the study site. As specified by the protocol, the percentage of participants negative for bilirubin, erythrocytes, ketones, leukocytes, nitrite and protein on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available urinalysis data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Percentage of Participants
  Bilirubin Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Bilirubin Day 28 | 100 | 100 | 100 | 100
  Bilirubin Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Bilirubin Day 56 | 100 | 100 | 100 | 100
  Erythrocytes Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Erythrocytes Day 28 | 85.7 | 100 | 90.9 | 71.4
  Erythrocytes Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Erythrocytes Day 56 | 100 | 100 | 100 | 85.7
  Ketones Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Ketones Day 28 | 92.9 | 100 | 100 | 100
  Ketones Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Ketones Day 56 | 100 | 100 | 100 | 100
  Leukocytes Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Leukocytes Day 28 | 92.9 | 100 | 100 | 100
  Leukocytes Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Leukocytes Day 56 | 100 | 100 | 100 | 100
  Nitrite Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Nitrite Day 28 | 100 | 100 | 100 | 100
  Nitrite Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Nitrite Day 56 | 100 | 100 | 100 | 100
  Protein Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Protein Day 28 | 100 | 92.9 | 100 | 100
  Protein Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Protein Day 56 | 100 | 100 | 81.8 | 100

19. Secondary Outcome: Laboratory Parameters (Urinalysis): Percentage of Participants Normal for Glucose and Urobilinogen on Days 28 and 56
Description: Urinalysis parameters were investigated in urine samples from participants by means of clinical laboratory assays and evaluated by the investigator. Glucose and urobilinogen were defined as normal by the local laboratory and reported at the study site. As specified by the protocol, the percentage of participants normal for glucose and urobilinogen on Day 28 (second dose) and Day 56 (follow-up assessment) was presented.
Time Frame: Day 28 and Day 56
Population: All randomized participants who received at least one dose of study treatment and had available urinalysis data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 8
Percentage of Participants
  Glucose Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Glucose Day 28 | 100 | 100 | 100 | 100
  Glucose Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Glucose Day 56 | 100 | 100 | 100 | 100
  Urobilinogen Day 28: number analyzed (Participants) | 14 | 14 | 11 | 7
  Urobilinogen Day 28 | 100 | 100 | 100 | 100
  Urobilinogen Day 56: number analyzed (Participants) | 14 | 14 | 11 | 7
  Urobilinogen Day 56 | 100 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: Up to 182 Days
Description: The analysis population included all randomized participants who received at least one dose of study treatment. Per protocol, adverse events were analyzed per treatment group but were not assessed with respect to individual vaccinations.
Arm/Group | Group A: V187 (High Dose) - V187 (High Dose) | Group B: V187 (Low Dose) - V187 (Low Dose) | Group C: V187 (High Dose) - Placebo | Group D: Placebo - Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 13/14 | 13/14 | 11/12 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: V187 (High Dose) - V187 (High Dose) (N=14) | Group B: V187 (Low Dose) - V187 (Low Dose) (N=14) | Group C: V187 (High Dose) - Placebo (N=12) | Group D: Placebo - Placebo (N=8)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: V187 (High Dose) - V187 (High Dose) (N=14) | Group B: V187 (Low Dose) - V187 (Low Dose) (N=14) | Group C: V187 (High Dose) - Placebo (N=12) | Group D: Placebo - Placebo (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (8) | 1 (2) | 1 (1) | 1 (3)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (6) | 3 (3) | 2 (5) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Injection site pain (General disorders) | 13 (31) | 9 (17) | 8 (10) | 2 (2)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 4 (5) | 2 (3) | 1 (2)
Oral herpes (Infections and infestations) | 1 (1) | 3 (3) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 5 (7) | 8 (14) | 3 (5)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators may not submit the results for publication or presentation without prior written permission of the sponsor. Authorship for any publication will be determined in mutual agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT04033068/Prot_SAP_000.pdf